CLINICAL TRIAL: NCT05202925
Title: Feasibility Study of a Musical Training Program in Improving the Neurocognitive Functioning of Children Surviving Brain Tumours
Brief Title: Musical Training Programme to Improve Neurocognitive Functioning of Children Surviving Brain Tumours
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Health and Medical Research Fund (Other Government)
Responsible Party: Principal Investigator, Dr Joyce Chung, Assistant Professor, School of Nursing, The Hong Kong Polytechnic University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HKCH-REC-2021-008
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Cancer Childhood; Brain Tumor
MeSH Terms: conditions — Neoplasms; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Musical Training (Experimental): All subjects in the intervention group will receive a weekly 45-minute lesson, one-to-one musical training for 52 weeks.
  Interventions: Other: Musical Training Program

INTERVENTIONS:
Other: Musical Training Program — a weekly 45-minute lesson, one-to-one musical training

SUMMARY:
We aim to conduct a feasibility study to determine the feasibility and suitability of implementing a musical training program for children surviving brain tumours. This study will demonstrate the feasibility of implementing a musical training program in improving the neurocognitive functioning of surviving brain tumours.

DETAILED DESCRIPTION:
Brain tumour is the second most common childhood cancer in Hong Kong. Evidence shows that cancer and its treatments have long-term and lasting adverse effects on the neurocognitive functioning of paediatric brain tumour survivors, including the impairment of intellectual development and deficits in attention, working memory, processing speed and executive functions. There has been an increase in the use of musical training to promote the neuro-rehabilitation of patients suffering from stroke and Parkinson's disease, and to improve reading skills and academic achievement in young poor readers, and to enhance children's cognitive development. We conducted a randomized controlled trial (RCT) from 2017 to 2018 to examine the effectiveness of musical training on psychological outcomes and quality of life in Chinese paediatric brain tumour survivors. The results showed that participants who received a weekly 45-min lesson on musical training for 52 weeks (intervention group) reported statistically significant fewer depressive symptoms, higher levels of self-esteem, and better quality of life than those who received placebo intervention (control group) at 12-month demonstrating the effectiveness of musical training intervention. Nevertheless, it is unclear whether musical training can also be used to improve neurocognitive functioning, in particular the attention, processing speed, and executive functions of children surviving brain tumours.

The overall aim of this proposed study will be to assess the feasibility of a musical training program in improving the neurocognitive functioning of children surviving brain tumours. The objectives of this feasibility study are as follows:

1. To ascertain the feasibility of recruitment and data collection in the outpatient clinic of the Hong Kong Children's Hospital;
2. To assess the response and retention rates of the study;
3. To examine the content of the proposed musical training program for its appropriateness, comprehensiveness and duration to the target participants;
4. To evaluate the appropriateness and feasibility of using various assessment tools in measuring the intelligence, attention, processing speed and executive functions of the paediatric brain tumour survivors; and
5. To assess any changes in neurocognitive functioning of children surviving brain tumours after receiving musical training for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. children who have completed cancer treatment at least 2 months previously;
2. aged between 7 and 16 years,
3. able to speak Cantonese and read Chinese, and
4. those who have not undertaken any musical training following their cancer diagnosis.

Exclusion Criteria:

1. those survivors with evidence of cancer recurrence or second malignancy in their medical records

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Recruitment rate of the study | at baseline before the start of the intervention
  the proportion of subjects who are eligible and invited and consent to participate.
Response rate of the study | at baseline and 12 months after starting the intervention
  The proportion of subjects who complete the questionnaires and assessments at baseline and 12 months after starting the intervention
Retention rate of the study | at baseline and 12 months after starting the intervention
  The proportion of subjects who complete the whole intervention from baseline to 12 months.

SECONDARY OUTCOMES:
Nonverbal intelligence scores of the subject | at baseline and 12 months after starting the intervention
  Measured by the Test of Nonverbal Intelligence, 4th edition (TONI-4)
Attention scores of the subject | at baseline and 12 months after starting the intervention
  Measured by the Digit Span
Processing speed scores of the subject | at baseline and 12 months after starting the intervention
  Measured by the Children's Color Trails Test (CCTT)
Executive functions scores of the subject | at baseline and 12 months after starting the intervention
  Measured by the Children's Color Trails Test (CCTT)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Chung, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Children's Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Chung JOK, Li WHC, Leung YD, Cheung TCK, Chiu SY, Pong MSY, Chan GCF. The feasibility, acceptability, and potential efficacy of a musical training program in promoting neuroplasticity among survivors of pediatric brain tumors: A cohort study. Eur J Oncol Nurs. 2025 Jun;76:102851. doi: 10.1016/j.ejon.2025.102851. Epub 2025 Feb 28. PMID 40043524